CLINICAL TRIAL: NCT01756131
Title: An Observer- and Subject-Blinded, Randomized, Placebo-Controlled, Single Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of Intramuscular and Subcutaneous Long Acting GSK1265744 in Healthy Subjects
Brief Title: A Single Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of Intramuscular and Subcutaneous Long Acting GSK1265744 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 114433; NCT01215006 (obsolete NCT alias)
Record Dates: First submitted 2011-09-01; First posted 2012-12-25 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-03

CONDITIONS: Infections, Human Immunodeficiency Virus and Herpesviridae
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — cabotegravir

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Cohort 1 (Experimental): 100 mg GSK1265744 injectable suspension or placebo, intramuscular dosing
  Interventions: Drug: GSK1265744 injectable suspension; Other: Placebo to match injectable suspension
- Cohort 2 (Experimental): 200 mg GSK1265744 injectable suspension or placebo, intramuscular dosing
  Interventions: Drug: GSK1265744 injectable suspension; Other: Placebo to match injectable suspension
- Cohort 3 (Experimental): 400 mg GSK1265744 injectable suspension or placebo, intramuscular dosing
  Interventions: Drug: GSK1265744 injectable suspension; Other: Placebo to match injectable suspension
- Cohort 4 (Experimental): 800 mg GSK1265744 injectable suspension or placebo, intramuscular dosing
  Interventions: Drug: GSK1265744 injectable suspension; Other: Placebo to match injectable suspension
- Cohort 5 (Experimental): 100 mg GSK1265744 injectable suspension or placebo, subcutaneous dosing
  Interventions: Other: Placebo to match injectable suspension
- Cohort 6 (Experimental): 200 mg GSK1265744 injectable suspension or placebo, subcutaneous dosing
  Interventions: Other: Placebo to match injectable suspension
- Cohort 7 (Experimental): 400 mg GSK1265744 injectable suspension or placebo, subcutaneous dosing
  Interventions: Drug: GSK1265744 injectable suspension
- Cohort 8 (Experimental): 400 mg GSK1265744 injectable suspension or placebo, intramuscular dosing
  Interventions: Drug: GSK1265744 injectable suspension
- Cohort 9 (Experimental): 400 mg GSK1265744 injectable suspension or placebo, intramuscular dosing
  Interventions: Drug: GSK1265744 injectable suspension

INTERVENTIONS:
Drug: GSK1265744 injectable suspension — 200 milligram per milliliter sterile solution for injection
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 7; Cohort 8; Cohort 9
Other: Placebo to match injectable suspension — placebo
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6

SUMMARY:
A single dose escalation study to determine the safety, tolerability, and pharmacokinetic profile of intramuscular and subcutaneous injections of GSK1265744 long acting parenteral (LAP) in healthy subjects. This study consists of a screening visit, a single injection, and follow-up evaluations for a minimum of 12 weeks following the injection.

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Females of childbearing potential with a negative pregnancy test (serum or urine) at screen and at Day -1, and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the investigational product is undetectable.
* Body weight greater than or equal to 50 kilograms (kg) for men and greater than or equal to 45 kg for women and body mass index (BMI) within the range 18.5-31.0 kilograms per meters squared (inclusive).
* Average QTcB or QTcF less than 450 milliseconds (msec); or QTc less than 480 msec in subjects with Bundle Branch Block.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* A positive pre-study Hepatitis B surface antigen, positive Hepatitis C antibody, or positive test for HIV antibody result within 3 months of screening
* High-risk behavior for Human Immunodeficiency Virus (HIV) infection including one of the following risk factors within six months before entering the study (day 1): Unprotected vaginal or anal sex with a known HIV infected person or a casual partner, engaged in sex work for money or drugs, acquired a sexually transmitted disease, high risk partner currently or in the previous six months.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation. If heparin is used during pharmacokinetics sampling, subjects with a history or sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* A positive pre-study drug screen.
* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of greater than 14 drinks for males or greater than 7 drinks for females.

* Unwilling to abstain from alcohol from 48 hours prior to admission to study site (Day -1) until discharge from clinic and for 48 hours prior to drawing clinical laboratory tests (Day 7, Day 14, Week 3, Week 4, Week 6, Week 8, Week 12, and follow-up [if necessary]).
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliters (mL) within a 56 day period
* Lactating females.
* The subject has an underlying skin disease or disorder (i.e. infection, inflammation, dermatitis, eczema, drug rash, drug allergy, psoriasis, food allergy, urticaria).
* The subject has a tattoo or other dermatological condition overlying the gluteus and/or abdominal region which may interfere with interpretation of injection site reactions.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, and direct bilirubin values above 1.5 times the upper limit of normal (isolated bilirubin greater than 1.5 times the upper limit of normal is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* The subject's systolic blood pressure is outside the range of 90-140 millimeters of mercury (mmHg), or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100 beats per minute (bpm) for female subjects or 45-100 bpm for male subjects.
* History of clinically significant cardiovascular disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
GSK1265744 safety and tolerability parameters including: the collection of adverse events | 12 weeks
Change from baseline values in clinical laboratory assessments | 12 weeks
Change from baseline for Electrocardiogram (ECG) assessments | 12 weeks
Change from baseline valuse in vital sign assessments (systolic and diastolic blood pressure and pulse rate) | 12 weeks
Composite of pharmacokinetic parameters: pre-dose and at 4, 8, 12 hours, Day 2, Days 3, 4, 5, 6, 7, Weeks 3, 4, 5, 6, 8, 12 and every 4 weeks until GSK1265744 is less than 0.10 or until 24 weeks | 12 weeks
  GSK1265744 pharmacokinetic parameters: area under the plasma concentration time curve from time zero to the last quantifiable time points (AUC(0-tau)), area under the plasma concentration time curve from time zero to infinity (AUC(0-infinity)), maximum observed concentration (Cmax), time to maximum observed concentration (tmax), apparent terminal phase half-life for LAP administration (t½), lambda z as a measure of absorption rate constant
GSK1265744 concentration at 1 month post-dose (C720 hours) | 4 weeks

SECONDARY OUTCOMES:
Composite of pharmacokinetic parameters: pre-dose and at 4, 8, 12 hours, Day 2, Days 3, 4, 5, 6, 7, Weeks 3, 4, 5, 6, 8, 12 and every 4 weeks until GSK1265744 is less than 0.10 or until 24 weeks. | 12 weeks
  GSK1265744 pharmacokinetic parameters: absorption lag time (tlag), apparent clearance (CL/F,LAP) following single dose administration, Percentage of AUC(0-infinity) obtained by extrapolation (AUC%ex)
Composite of pharmacokinetic parameters for dose proportionality: pre-dose and at 4, 8, 12 hours, Day 2, Days 3, 4, 5, 6, 7, Weeks 3, 4, 5, 6, 8, 12 and every 4 weeks until GSK1265744 is less than 0.10 or until 24 weeks | 12 weeks
  GSK1265744 following single dose administration at different doses for the assessment of dose proportionality: AUC(0-infinity), AUC(0-tau), Cmax
GSK1265744 C720 hours following single dose administration at different doses for the assessment of dose proportionality | 12 weeks
GSK1265744 concentrations in cervicovaginal fluid (CVF), cervical tissue (CT), vaginal tissue (VT), rectal tissue (RT), and blood plasma and ratio of CVF, CT, VT, and RT concentration to blood plasma | Cohort 8 at week 2 and week 8; Cohort 9 at week 4 and week 12
  Cohort 8 at week 2 and week 8; Cohort 9 at week 4 and week 12

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare